CLINICAL TRIAL: NCT04624451
Title: Evaluation of Intravenous Dalbavancin for Treatment of Peritonitis in Peritoneal Dialysis Patients
Brief Title: Evaluation of Intravenous Dalbavancin for Peritonitis
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1731
Record Dates: First submitted 2020-07-09; First posted 2020-11-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Peritonitis; Peritonitis Bacterial
MeSH Terms: conditions — Peritonitis | interventions — dalbavancin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Dalbavancin — Dalbavancin 1500 mg intravenously x 1 dose

SUMMARY:
This study evaluates the use of Dalbavancin 1500 mg IV x 1 dose for treating patients with gram positive peritonitis in patients requiring peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

Patients > 18 years of age actively receiving peritoneal dialysis diagnosed with a gram + peritonitis determined to be a good candidate for dalbavancin treatment by the attending nephrology attending.

Exclusion Criteria:

Patients with contraindications to dalbavancin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently receiving peritoneal dialysis that are found to have bacterial peritonitis
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical cure | 14 days
  resolution of signs and symptoms (e.g. abdominal pain), bacterial eradication, reduction in clinical markers (e.g. peritoneal fluid findings, CRP, etc), and return of peritoneal dialysis functionality
Clinical cure | 28 days
  resolution of signs and symptoms (e.g. abdominal pain), bacterial eradication, reduction in clinical markers (e.g. peritoneal fluid findings, CRP, etc), and return of peritoneal dialysis functionality

SECONDARY OUTCOMES:
Treatment emergent adverse events | 14 days
  Occurrence of any adverse events
Treatment emergent adverse events | 28 days
  Occurrence of any adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Matre ET, Teitelbaum I, Kiser TH. Intravenous and Intraperitoneal Pharmacokinetics of Dalbavancin in Peritoneal Dialysis Patients. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02089-19. doi: 10.1128/AAC.02089-19. Print 2020 Apr 21. PMID 32122898